CLINICAL TRIAL: NCT02806024
Title: Perioperative Administration of Tranexamic Acid for Placenta Previa and Accreta Study (TAPPAS): A Randomized, Placebo-controlled Double Blind Trial
Brief Title: Perioperative Administration of Tranexamic Acid for Placenta Previa and Accreta Study
Acronym: TAPPAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Central California Faculty Medical Group (Other)
Responsible Party: Principal Investigator, Mallory Kremer, Principle Investigator, Clinical Instructor, University of California, San Francisco
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 2016036
Record Dates: First submitted 2016-06-10; First posted 2016-06-20 (Estimated); Results first posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Placenta Accreta; Postpartum Hemorrhage; Cesarean Section; Tranexamic Acid
MeSH Terms: conditions — Placenta Accreta; Postpartum Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment Arm (Tranexamic Acid, or TXA) (Experimental): Patients will be randomized to treatment or placebo arms preoperatively. In our treatment arm of pregnant patients with suspected placenta accreta or at high risk for placenta accreta, patients will receive 1 gram intravenous TXA administered over 10 minutes immediately after delivery of the infant. The drug will be prepared and ready to hang at the beginning of the case. The study drug will be administered only once.
  Interventions: Drug: Tranexamic Acid
- Placebo Arm (Placebo Comparator): Patients will be randomized to treatment or placebo arms preoperatively. In our placebo arm of pregnant patients with suspected placenta accreta, patients will receive plain normal saline in a 50 cc bag identical to the preparation of study drug immediately after delivery of the infant.
  Interventions: Drug: Placebo Drug

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Treatment Arm (Tranexamic Acid, or TXA)
Drug: Placebo Drug — 50 cc Normal Saline IV
  Arms: Placebo Arm

SUMMARY:
The purpose of this pilot study is to determine if intravenous tranexamic acid (TXA) is effective for reducing blood loss during high risk surgical procedures related to placenta previa and placenta accreta. TXA is currently used in other types of surgery for patients who are expected to have a large blood loss, such as orthopedic or open heart surgery.

DETAILED DESCRIPTION:
To date, no novel or pharmacologic methods of reducing blood loss have been described for women at risk for placenta accreta. Intravenous tranexamic acid (TXA), a drug with anti-fibrinolytic activity, is routinely used in elective orthopedic and cardiac surgery to reduce blood loss. Intravenous tranexamic acid is currently FDA approved for use in patients undergoing cardiac surgery or total knee arthroplasty or total hip arthroplasty to reduce peri- and post-operative blood loss and to reduce the need for blood transfusion. There has been growing interest in the application of tranexamic acid in obstetrics and gynecology. In multiple international studies, intravenous TXA has been shown to significantly reduce blood loss when given prophylactically with cesarean delivery or vaginal delivery without an increase in morbidity from adverse thrombotic events. TXA has not been studied in the particular population of patients requiring cesarean hysterectomy for placenta previa or accreta. This inexpensive, low risk medication has potential to greatly reduce perioperative morbidity and cost when used in a high risk obstetrical population.

ELIGIBILITY:
Inclusion Criteria:

* English and Spanish speaking pregnant women
* Any order pregnancy (singleton, twin gestation, etc)
* Suspected accreta based on ultrasound or MRI imaging studies
* All women evaluated for placenta accreta and deemed to be high risk for this disease (≥40% risk), meaning women diagnosed with a placenta previa and greater than or equal to 2 prior c-sections

Exclusion Criteria:

* Women less than 18 years of age
* Women with a personal history of venous or arterial thrombosis (deep vein thrombosis, pulmonary embolism, myocardial infarction, or stroke
* Women with a personal history of a high risk clotting disorder, such as anti-phospholipid syndrome
* Women who do not have a good understanding of either English or Spanish will be excluded.
* Women with defective color vision (color-blindness)

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Community Regional Medical Center, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Novikova N, Hofmeyr GJ, Cluver C. Tranexamic acid for preventing postpartum haemorrhage. Cochrane Database Syst Rev. 2015 Jun 16;2015(6):CD007872. doi: 10.1002/14651858.CD007872.pub3. PMID 26079202
- [Background] Silver RM, Landon MB, Rouse DJ, Leveno KJ, Spong CY, Thom EA, Moawad AH, Caritis SN, Harper M, Wapner RJ, Sorokin Y, Miodovnik M, Carpenter M, Peaceman AM, O'Sullivan MJ, Sibai B, Langer O, Thorp JM, Ramin SM, Mercer BM; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Maternal morbidity associated with multiple repeat cesarean deliveries. Obstet Gynecol. 2006 Jun;107(6):1226-32. doi: 10.1097/01.AOG.0000219750.79480.84. PMID 16738145
- [Background] Abdel-Aleem H, Alhusaini TK, Abdel-Aleem MA, Menoufy M, Gulmezoglu AM. Effectiveness of tranexamic acid on blood loss in patients undergoing elective cesarean section: randomized clinical trial. J Matern Fetal Neonatal Med. 2013 Nov;26(17):1705-9. doi: 10.3109/14767058.2013.794210. Epub 2013 May 10. PMID 23574458

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were women with suspicion of morbidly adherent placenta (accreta) on imaging, or women with placenta previa and two or more cesareans (CS).
Pre-assignment Details: One patient was excluded from the study after consenting to participate, but before delivery. Two consented patients delivered at night, and were unable to be randomized.
Groups:
- Treatment Arm (Tranexamic Acid, or TXA): Patients will be randomized to treatment or placebo arms preoperatively. In our treatment arm of pregnant patients with suspected placenta accreta or at high risk for placenta accreta, patients will receive 1 gram intravenous TXA administered over 10 minutes immediately after delivery of the infant. The drug will be prepared and ready to hang at the beginning of the case. The study drug will be administered only once.
  Tranexamic Acid
Period: Overall Study
Arm/Group | Treatment Arm (Tranexamic Acid, or TXA) | Placebo Arm
Started | 7 | 7
Completed | 6 | 5
Not Completed | 1 | 2
Not completed — Night Delivery | 1 | 1
Not completed — DVT during antepartum admission | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm (Tranexamic Acid, or TXA) | Placebo Arm | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (2.2) | 31.0 (7.9) | 30.2 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 4 | 3 | 7
  Asian | 1 | 0 | 1
  Black | 0 | 1 | 1
  White | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Estimated Blood Loss (EBL)
Description: EBL is estimated by the surgeon and anesthesia team at the completion of the surgery (cesarean delivery &/or cesarean hysterectomy).
Time Frame: 1-3 hours (will be determined at the completion of the surgery).
Population: Mean estimated blood loss (EBL) was calculated as below.
Measure: Mean (Standard Deviation); unit: cc
Arm/Group | Treatment Arm (Tranexamic Acid, or TXA) | Placebo Arm
Number analyzed (Participants) | 6 | 5
cc | 3116 (3947) | 9420 (12474)

2. Secondary Outcome: Blood Transfusion (Number of Units Transfused) Intraoperatively
Description: Total number of units of blood transfused (whole blood, platelets, cryoprecipitate, and fresh frozen plasma) intra-operatively is a secondary outcome.
Time Frame: Pulled from operative note, completed by the time of discharge.
Population: The mean pRBCs units given intraoperatively is presented in the table below.
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Treatment Arm (Tranexamic Acid, or TXA) | Placebo Arm
Number analyzed (Participants) | 6 | 5
units | 5.2 (8) | 17.6 (25)

ADVERSE EVENTS:
Time Frame: Enrollment to 6 weeks post partum.
Description: Patients were seen for routine post partum care and chart review was performed to glean adverse events from their hospital stay for delivery.
Arm/Group | Treatment Arm (Tranexamic Acid, or TXA) | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 4/6 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (Tranexamic Acid, or TXA) (N=6) | Placebo Arm (N=5)
DVT / PE (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (Tranexamic Acid, or TXA) (N=6) | Placebo Arm (N=5)
Urinary tract injury during surgery (cystotomy or ureter injury) (Renal and urinary disorders) | 2 (2) | 2 (2)
Wound infection (Surgical and medical procedures) | 1 (1) | 1 (1) — Post operative wound seroma
IR balloon complication (Surgical and medical procedures) | 1 (1) | 0 (0) — Interventional radiology balloon complication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-09-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT02806024/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-06-04): https://cdn.clinicaltrials.gov/large-docs/24/NCT02806024/Prot_SAP_001.pdf